CLINICAL TRIAL: NCT06896032
Title: Effect of Retro-walking Versus Forward-walking Training Using Underwater Treadmill on Pain and Function in Patients With Knee Osteoarthritis
Brief Title: Retro-walking Versus Forward-walking Training Using Underwater Treadmill in Patients With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan Atwa Said (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Nourhan Atwa Said, physical therapist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005428
Record Dates: First submitted 2025-02-22; First posted 2025-03-26 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-03

CONDITIONS: Knee Osteoarthritis (Knee OA); Osteoarthritis
Keywords: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: Retro walking and forward walking training exercise
Who Masked: Investigator, Outcomes Assessor
Masking Description: Opaque sealed envelope
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- group A (experimental1) (Experimental): forward walking group
  Interventions: Other: physical therapy intervention
- group B (experimental 2) (Experimental): retro walking group
  Interventions: Other: physical therapy intervention
- group c (Other): control group
  Interventions: Other: physical therapy intervention

INTERVENTIONS:
Other: physical therapy intervention — retro-walking and forward-walking underwater treadmill training
  Other Names: hydro therapy; aquatic therapy

SUMMARY:
The purpose of this study Will investigate and compare the effects of retro-walking and forward-walking underwater treadmill training on pain, function and ROM in subjects with chronic knee OA

DETAILED DESCRIPTION:
In the current study, Sixty subjects from both genders, the dominant side only will be involved. They will be divided in to three equal groups: group A (experimental1), group B (experimental 2), group C (control), they will be signed a consent form to share in this study which aimed to investigate the effects of retro-walking and forward-walking underwater treadmill training on pain, function and ROM in subjects with chronic knee OA

ELIGIBILITY:
Inclusion Criteria:

1. 60 patients with chronic knee OA.
2. Age ranges from 40-60 years old of both genders.
3. body mass index (BMI) 25- 35kg/m2.
4. The degree of osteoarthritis was mild or moderate and have a Kellgren- Lawrence radiographic grade of of1-3.
5. unilateral knee osteoarthritis involvement.

Exclusion Criteria:

1. hydrophobia.
2. pregnancy.
3. infection.
4. psychiatric disorder.
5. haemorrhagic diathesis.
6. cardiac pacemaker.
7. all Subjects with deformity of hip, knee & ankle.
8. any CNS or PNS involvement.
9. recent steroidal or intraarticular injections (3 months).
10. systemic inflammatory disease and bone malignancy.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | up to three monthes
  Pain intensity will be measured by visual analog scale (VAS. ). It is line with worst pain at one end and no pain at the other end
knee disability | up to three months
  knee disablity will be measured by The Western Ontario and McMaster Universities osteoarthritis index. The WOMAC is a self-administered instrument containing 24 items measuring 3 subscales: physical function (17 items), pain (5 items), and stiffness (2 items).Scores range from 0 to 96 for the total WOMAC where 0 represents the best health status and 96 the worst possible status.

SECONDARY OUTCOMES:
knee range of motion | up to three months
  knee joint rang of motion will be measured by goniometer

CONTACTS AND LOCATIONS:
Locations (1):
- cairo U, Cairo, Cairo Governorate, Egypt